CLINICAL TRIAL: NCT04639050
Title: A Phase Ib/IIa, Randomized, Double Blind, Placebo-Controlled, Multiple Ascending Dose, Parallel-Group Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of RO7126209 Following Intravenous Infusion in Patients With Prodromal or Mild to Moderate Alzheimer's Disease
Brief Title: Brainshuttle AD: A Multiple Ascending Dose Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of RO7126209 Following Intravenous Infusion in Participants With Prodromal or Mild to Moderate Alzheimer's Disease
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BP42155; 2020-002477-98 (EudraCT Number); 2023-509678-52-00 (Other: EU Trial Number)
Record Dates: First submitted 2020-11-17; First posted 2020-11-20 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Alzheimers Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (19):
- Part 1 (Dose Finding) Cohort 1: Dose Level 1 of RO7126209 (Experimental): Participants will receive multiple doses of RO7126209 at dose level 1 once every 4 weeks (Q4W) for 28 weeks followed by a 28-week safety follow-up period.
  Interventions: Drug: RO7126209
- Part 1 (Dose Finding) Cohort 1: Placebo (Placebo Comparator): Participants will receive matching placebo to dose level 1 Q4W for 28 weeks followed by a 28-week safety follow-up period.
  Interventions: Drug: Placebo
- Part 1 (Dose Finding) Cohort 2: Dose Level 2 of RO7126209 (Experimental): Participants will receive multiple doses of RO7126209 at dose level 2, Q4W, for 28 weeks followed by a 28-week safety follow-up period.
  Interventions: Drug: RO7126209
- Part 1 (Dose Finding) Cohort 2: Placebo (Placebo Comparator): Participants will receive matching placebo to dose level 2, Q4W, for 28 weeks followed by a 28-week safety follow-up period.
  Interventions: Drug: Placebo
- Part 1 (Dose Finding) Cohort 3: Dose Level 3 of RO7126209 (Experimental): Participants will receive multiple doses of RO7126209 at dose level 3, Q4W, for 28 weeks followed by a 28-week safety follow-up period.
  Interventions: Drug: RO7126209
- Part 1 (Dose Finding) Cohort 3: Placebo (Placebo Comparator): Participants will receive matching placebo to dose level 3, Q4W, for 28 weeks followed by a 28-week safety follow-up period.
  Interventions: Drug: Placebo
- Part 1 (Dose Finding) Cohort 4: Dose Level 4 of RO7126209 (Experimental): Participants will receive multiple doses of RO7126209 at dose level 4, Q4W, for 28 weeks followed by a 28-week safety follow-up period.
  Interventions: Drug: RO7126209
- Part 1 (Dose Finding) Cohort 4: Placebo (Placebo Comparator): Participants will receive matching placebo to dose level 4, Q4W, for 28 weeks followed by a 28-week safety follow-up period.
  Interventions: Drug: Placebo
- Part 1 (Dose Finding) Cohort 5: Dose Level 5 of RO7126209 (Experimental): Participants will receive a total of 2 doses of RO7126209 at dose level 5 Q4W, for 28 weeks followed by an 8-week safety follow-up period.
  Interventions: Drug: RO7126209
- Part 1 (Dose Finding) Cohort 5: Placebo (Placebo Comparator): Participants will receive a total of 2 doses of matching placebo to dose level 5 Q4W, for 28 weeks followed by an 8-week safety follow-up period.
  Interventions: Drug: Placebo
- Part 2 (Expansion) Cohort 1: Dose Level 3 of RO7126209 (Experimental): Participants will receive multiple doses of RO7126209 at dose level 3, Q4W, for 28 weeks followed by a 28-week safety follow-up period.
  Interventions: Drug: RO7126209
- Part 2 (Expansion) Cohort 1: Placebo (Placebo Comparator): Participants will receive matching placebo to dose level 3, Q4W, for 28 weeks followed by a 28-week safety follow-up period.
  Interventions: Drug: Placebo
- Part 2 (Expansion) Cohort 2: Dose Level 4 of RO7126209 (Experimental): Participants will receive multiple doses of RO7126209 at dose level 4, Q4W, for 28 weeks followed by a 28-week safety follow-up period.
  Interventions: Drug: RO7126209
- Part 2 (Expansion) Cohort 2: Placebo (Placebo Comparator): Participants will receive matching placebo to dose level 4, Q4W, for 28 weeks followed by a 28-week safety follow-up period.
  Interventions: Drug: Placebo
- Part 2 (Expansion) Cohort 3: Dose Level 5 of RO7126209 (Experimental): Participants will receive a total of 2 doses of RO7126209 at dose level 5, Q4W, for 28 weeks followed by an 8-week safety follow-up period.
  Interventions: Drug: RO7126209
- Part 2 (Expansion) Cohort 3: Placebo (Placebo Comparator): Participants will receive a total of 2 doses of matching placebo to dose level 5, Q4W, for 28 weeks followed by an 8-week safety follow-up period.
  Interventions: Drug: Placebo
- Part 3 (Dose/Frequency/Pharmacodynamic (PD) Relationship): Dose Level 1: RO7126209 (Experimental): Participants will receive multiple doses of RO7126209 in an open-label treatment period at dose level 1, Q4W, for 24 weeks followed by a 28-week safety follow-up period.
  Interventions: Drug: RO7126209
- Part 3 Dose/Frequency/PD Relationship: Dose Level 2: RO7126209 (Experimental): Participants will receive multiple doses of RO7126209 in an open-label treatment period at dose level 2, Q12W, for 24 weeks followed by a 28-week safety follow-up period.
  Interventions: Drug: RO7126209
- Part 4: Open Label Extension (OLE) (Experimental): Participants who completed Part 1, 2, or 3 will receive RO7126209 for a maximum of 205 weeks.
  Interventions: Drug: RO7126209

INTERVENTIONS:
Drug: RO7126209 — RO7126209 will be administered intravenously as specified in each treatment arm.
  Other Names: Trontinemab; RG6102
  Arms: Part 1 (Dose Finding) Cohort 1: Dose Level 1 of RO7126209; Part 1 (Dose Finding) Cohort 2: Dose Level 2 of RO7126209; Part 1 (Dose Finding) Cohort 3: Dose Level 3 of RO7126209; Part 1 (Dose Finding) Cohort 4: Dose Level 4 of RO7126209; Part 1 (Dose Finding) Cohort 5: Dose Level 5 of RO7126209; Part 2 (Expansion) Cohort 1: Dose Level 3 of RO7126209; Part 2 (Expansion) Cohort 2: Dose Level 4 of RO7126209; Part 2 (Expansion) Cohort 3: Dose Level 5 of RO7126209; Part 3 (Dose/Frequency/Pharmacodynamic (PD) Relationship): Dose Level 1: RO7126209; Part 3 Dose/Frequency/PD Relationship: Dose Level 2: RO7126209; Part 4: Open Label Extension (OLE)
Drug: Placebo — RO7126209-matching placebo will be administered intravenously as specified in each treatment arm.
  Other Names: RO727-5887, F01-01
  Arms: Part 1 (Dose Finding) Cohort 1: Placebo; Part 1 (Dose Finding) Cohort 2: Placebo; Part 1 (Dose Finding) Cohort 3: Placebo; Part 1 (Dose Finding) Cohort 4: Placebo; Part 1 (Dose Finding) Cohort 5: Placebo; Part 2 (Expansion) Cohort 1: Placebo; Part 2 (Expansion) Cohort 2: Placebo; Part 2 (Expansion) Cohort 3: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, immunogenicity, pharmacokinetics, and pharmacodynamics of multiple-ascending intravenous (IV) doses of RO7126209 in participants with prodromal or mild to moderate Alzheimer's disease (AD), who are amyloid positive based on amyloid positron emission tomography (PET) scan.

ELIGIBILITY:
Key inclusion criteria for part 1, 2 and 3:

* Ability to provide written consent signed by the participant
* Availability of a person (referred to as the "study partner") who: consents to participate throughout the duration of study, in the Investigator's judgment, has frequent and sufficient contact with the participant, is fluent in the language of the tests used at the study site
* Willingness and ability to complete all aspects of the study (including magnetic resonance imaging [MRI], lumbar puncture, clinical genotyping, and positron emission tomography [PET] imaging)
* Capable of completing assessments either alone or with the help of the study partner
* Adequate visual and auditory acuity, in the Investigator's judgment, sufficient to perform the neuropsychological testing (eye glasses and hearing aids are permitted)
* Probable mild to moderate AD dementia (consistent with National Institute on Aging-Alzheimer's Association [NIA-AA] core clinical criteria for probable AD dementia) or prodromal AD (consistent with the NIA-AA diagnostic criteria and guidelines for mild cognitive impairment due to AD)
* Screening Mini-Mental State Examination (MMSE) score of 18 to 28 points, inclusive, within 84 days before baseline
* Clinical Dementia Rating-Global Score (CDR-GS) of 0.5, 1, or 2 within 84 days before baseline
* Positive amyloid PET scan (cut-off: >50 Centiloid units) within 12 months before baseline
* In case of treatment with symptomatic AD medications, dosing regimen must be stable for at least 8 weeks prior to baseline and until randomization
* Agreement not to donate blood or blood products for transfusion for the duration of the study and for 1 year after final dose of study drug
* Agreement not to participate in other research studies for the duration of this study
* Agree to apolipoprotein E (APOE) genotyping

Inclusion criteria for Part 4:

- Completed the treatment period in Part 1, Part 2, or Part 3 of the study

Key exclusion criteria for part 1, 2 and 3:

* Any evidence of other relevant neurological condition, including other (non-AD) neurodegenerative and neuropsychiatric conditions, neurovascular brain disorders, seizure disorders, inflammatory and infectious disorders of the central nervous system, trauma and delirium, among several others
* Other relevant medical conditions including significant hematological diseases, any clinically significant ophthalmologic diseases, decreased visual acuity in either eye, with a BCVA letter score of less than 20 letters on the Early Treatment Diabetic Retinopathy Study (ETDRS) chart or the Snellen equivalent of 20/400 if the ETDRS chart is not used
* Clinically significant cardiovascular diseases, chronic kidney disease, confirmed and unexplained impaired hepatic function, abnormal thyroid function, among several others
* History of hypersensitivity to biologic agents or any of the excipients in the formulation
* Clinically significant abnormalities (as judged by the Investigator) in laboratory test results (including complete blood count, chemistry panel, routine cerebrospinal fluid [CSF] parameters and urinalysis)
* MRI exclusion criteria: >2 lacunar infarcts (including lacunar infarcts in the cerebellum), any territorial infarct >1 cm^3, any white matter lesion that corresponds to an overall Fazekas score of 3 that requires at least one confluent hyperintense lesion on the fluid-attenuated inversion recovery (FLAIR) sequence, which is ≥20 mm in any dimension
* More than 4 microhemorrhages on MRI and/or presence of any focal area of leptomeningeal hemosiderosis based on the review performed by the central MRI reader prior to randomization
* Presence of any other significant cerebral abnormalities, including amyloid-related imaging abnormality-edema/effusion (ARIA-E), as assessed on MRI
* Inability to tolerate MRI procedures or contraindication to MRI
* Inability to undergo ophthalmological assessments
* Contraindication to lumbar puncture
* Contraindication to having a PET scan

Exclusion criteria for Part 4:

* Prematurely discontinued from the treatment period for study (i.e., before the start of the follow-up period of Part 1, Part 2, or Part 3) for any reason or meeting discontinuation criteria before the baseline visit of Part 4.
* Received any active investigational treatment other than RO7126209 during or since completion of Part 1, Part 2 or Part 3
* Any passive immunotherapy (immunoglobulin) since completion of Part 1, Part 2, or Part 3 that is meant to prevent or postpone cognitive decline.
* Use of anti-coagulation medications - Evidence of ongoing ARIA-E. In this case participant may enroll into Part 4 once the ARIA-E is resolved - Evidence of ongoing infusion-related reaction (IRR) or hypersensitivity reaction. In this case participant may enroll into Part 4 once the IRR is resolved.
* MRI evidence of any of the following at OLE baseline: evidence of ongoing ARIA-E, any ARIA-H (leptomeningeal hemosiderosis or microhemorrhages) that would require permanent discontinuation of study treatment, > 2 lacunar infarcts, Any territorial infarct > 1 cm^3, any white matter lesion that corresponds to an overall Fazekas score of 3 that requires at least one confluent hyperintense lesion on the FLAIR sequence, which is ≥ 20 mm in any dimension
* Any drop in hemoglobin of > 20% compared to predose on Day 1 or hemoglobin value below 10 g/dL

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2030-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Part 1, 2, 3, and 4: Percentage of Participants With Adverse Events (AEs) | Part 1 and 2: Up to approximately 56 weeks; Part 3: Up to approximately 52 weeks; Part 4: Up to approximately 233 weeks
Part 3: Change From Baseline in Brain Amyloid Load as Measured by Amyloid Positron Emission Tomography (PET) Scan | Up to approximately 24 weeks

SECONDARY OUTCOMES:
Part 1, 2, and 4: Change From Baseline in Brain Amyloid Load as Measured by Amyloid PET Scan | Part 1 and 2: Up to approximately 28 weeks; Part 4: Up to approximately 205 weeks
Part 1, 2, 3, and 4: Plasma Concentration of RO7126209 | Part 1 and 2: Up to approximately 32 weeks; Part 3: Up to approximately 24 weeks; Part 4: Up to approximately 209 weeks
Part 1, 2, 3, and 4: Cerebral Spinal Fluid (CSF) Concentration of RO7126209 | Part 1 and 2: Up to approximately 25 weeks; Part 3: Up to approximately 21 weeks; Part 4: Up to approximately 205 weeks
Part 1, 2, 3, and 4: Number of Participants With Anti-Drug Antibodies (ADAs) to RO7126209 | Part 1 and 2: Up to approximately 56 weeks; Part 3: Up to approximately 52 weeks; Part 4: Up to approximately 233 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (41):
- United States (17):
  - JEM Research LLC, Atlantis, Florida
  - K2 Medical Research-Winter Garden, Clermont, Florida
  - K2 Medical Research - The Villages, Lady Lake, Florida
  - K2 Medical Research, LLC, Maitland, Florida
  - Optimus U Corp, Miami, Florida
  - Charter Research - Winter Park/Orlando, Orlando, Florida
  - Advent Health Orlando, Orlando, Florida
  - Alzheimer's Research and Treatment Center, Stuart, Florida
  - Charter Research - Lady Lake/The Villages, The Villages, Florida
  - Alzheimer?s Research and Treatment Center, Wellington, Florida
  - Conquest Research, LLC, Winter Park, Florida
  - Alzheimer's Research and Treatment Center - Columbus, Columbus, Georgia
  - Center for Advanced Research & Education, Gainesville, Georgia
  - Quest Research Institute, Farmington Hills, Michigan
  - Summit Research Network Inc., Portland, Oregon
  - Abington Neurological Associates, Abington, Pennsylvania
  - Kerwin Research Center, LLC, Dallas, Texas
- Australia (2):
  - Heidelberg Repatriation Hospital, Heidelberg West, Victoria
  - Alfred Hospital, Melbourne, Victoria
- Canada (2):
  - Richmond Clinical Trials, Richmond, British Columbia
  - Toronto Memory Program, Toronto, Ontario
- Chile (2):
  - Centro de Investigación Clínica UC-CICUC, Santiago
  - Hospital Clinico Univ de Chile, Santiago
- Japan (6):
  - Yokohama City Minato Red Cross Hospital, Kanagawa
  - Koseikai Takeda Hospital, Kyoto
  - National Hospital Organization Utano National Hospital, Kyoto
  - Keio University Hospital, Tokyo
  - Tokyo Metropolitan Geriatric Hospital, Tokyo
  - Federation of National Public Service Personnel Mutual Aid Associations Tachikawa Hospital, Tokyo
- Poland (2):
  - Osrodek Badan Klinicznych Euromedis, Szczecin
  - NZOZ WCA, Wroc?aw
- South Korea (2):
  - Inha University Hospital, Incheon
  - Samsung Medical Center, Seoul
- Spain (7):
  - Hospital General De Catalunya, Sant Cugat del Vallès, Barcelona
  - Policlínica Guipuzcoa, Donostia / San Sebastian, Guipuzcoa
  - Fundación ACE, Barcelona
  - Hospital Clinic i Provincial, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Dr. Peset, Valencia
  - Hospital Universitario la Fe, Valencia
- UCL Institute of Neurology, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing